CLINICAL TRIAL: NCT01918722
Title: Clinical Re-evaluation of Removing Blood Stasis Therapy of Herbal Medicine in Treating Acute Cerebral Hemorrhage Safety
Brief Title: Clinical Re-evaluation of Removing Blood Stasis Therapy in Treating Acute Cerebral Hemorrhage Safety and Efficacy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JDZX2012074; JDZX2012074 (Other Grant/Funding Number: China national clinical study base project of TCM)
Record Dates: First submitted 2013-04-18; First posted 2013-08-08 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Intracerebral Hemorrhage
Keywords: Activating blood stagnation and expelling blood stasis; Hematoma enlargement; herbal medicine; traditional chinese medicine; random clinical trial
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ICH-1 (Experimental): herbal medicine with Hirudo, Tabanus,8 herbals, promote blood circulation function
  Interventions: Drug: ICH-1(herbal medicine with Hirudo, Tabanus)
- ICH-2 (Active Comparator): herbal medicine without Hirudo, Tabanus,Only 6 herbals
  Interventions: Drug: ICH-2(herbal medicine without Hirudo, Tabanus)
- placebo herbal medicine (Placebo Comparator): Placebo ：granula，dose twice a day by Oral or nasogastric tube for 10 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ICH-1(herbal medicine with Hirudo, Tabanus) — 8herbals (with 2 herbals of Activating blood stagnation and expelling blood stasis herbs) one dose, bid, for 10 days
  Other Names: PXZY
  Arms: ICH-1
Drug: placebo — placebo herbal medicine, one dose,bid, for 10 days
  Other Names: pxzyp
  Arms: placebo herbal medicine
Drug: ICH-2(herbal medicine without Hirudo, Tabanus) — (6herbals, without 2 herbals of promoting blood stasis) one dose, bid, for 10 days
  Other Names: NPXZY
  Arms: ICH-2

SUMMARY:
In order to investigate the time window of acute intracerebral hemorrhage(AICH) by "Blood Activating and Stasis Dispersing" therapy and to verify traditional methods if it would influence or enlarge the brain hematoma, test is made by random double-blind controlled. Patients are classified to （0-6h）and (6-72h) teams. Herbs is separated too. The period of the therapy lasts two weeks, and the follow up should last three months. The main indexes are mortality rate, disability rate and the brain hematoma situation. The review is made by the reference to (NIHSS),(GCS) and so on. So, the window time is determined through this test.

DETAILED DESCRIPTION:
objective: to investigate the safety and effect of acute cerebral hemorrhage treated with "Blood Activating and Stasis Dispersing" therapy and to verify the traditional methods can influence the brain hematoma enlargement or not.

Methods: from 2013.8 to 2015.12, 360 cases of AICH will be included in 13 research centers. Patients are randomly into 3 groups within 6hrs from onset,such as, group A, blood activating herbal medicine (8 herbals), Group B, herbal medicine without blood activating herbal(6 herbals), Group C, placebo for 10days. All the patients will be treated according AHA guideline of AICH. All patients will be set to the CT at the onset, 24h later and 10-14days after treatment. So the rate of enlargement of brain hematoma in the 72h later, mortality rate in the two weeks and the disability rate in the 90 days can be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* no younger than 18 yrs
* acute cerebral hemorrhage confirmed by brain CT scan
* within 6 hours from onset
* GCS≥6
* Sign the informed consent form

Exclusion Criteria:

* Tests have confirmed that cerebral hemorrhage caused by brain tumor, blood diseases, cerebrovascular malformation (anomaly) or aneurysm, etc;
* patients with Severe heart, liver and renal insufficiency.
* Intolerance to traditional Chinese medicine (TCM), allergic constitution.
* patients with severe cerebral hernia in the early onset
* Compliance is poor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Hematoma enlargement | 24hrs, 10-14days

SECONDARY OUTCOMES:
fatality rate | 3 month
modified rankin scale | 3 months
National Institute of Health of stroke scale | 10-14days, 90days

CONTACTS AND LOCATIONS:
Overall Officials: Jianwen m Guo, doctor, Principal Investigator — Guangdong Province Hospital of Tradtional Chinese Medicine
Locations (15):
- China (15):
  - Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Guangzhou Hospital of Integrated traditional and west medicine, Guangzhou, Guangdong
  - Panyu Hospital of Chinese Medicine, Guangzhou, Guangdong
  - Boluo County People's Hospital, Huizhou, Guangdong
  - Jiangmen Wuyi Traditional Chinese Medicine Hospital, Jiangmen, Guangdong
  - The hospital of Chinese Medicine of Conghua City, Jiekou, Guangdong
  - Lianjiang People's hospital, Lianjiang, Guangdong
  - Zengcheng City Hospital of traditional Chinese Medicine, Licheng, Guangdong
  - Boji-affiliated Hospital of Sun Yat-sen University, Licheng, Guangdong
  - Yangjiang Hospital of Traditional Chinese Medicine, Yangjiang, Guangdong
  - 1st people's hospital of Yueyang city, Yueyang, Hunan
  - Shenyang No.2 traditional Chinese medical hospital, Shenyang, Liaoning
  - Liaocheng City People's Hospital, Liaocheng, Shandong
  - Shouguang City People's Hospital, Shouguang, Shandong

IPD SHARING:
Plan to Share IPD: Yes
The study has recruited 278 subjects by so far

REFERENCES:
- [Derived] Zeng L, Tang G, Wang J, Zhong J, Xia Z, Li J, Chen G, Zhang Y, Luo S, Huang G, Zhao Q, Wan Y, Chen C, Zhu K, Qiao H, Wang J, Huang T, Liu X, Zhang Q, Lin R, Li H, Gong B, Chen X, Zhou Y, Wen Z, Guo J. Safety and efficacy of herbal medicine for acute intracerebral hemorrhage (CRRICH): a multicentre randomised controlled trial. BMJ Open. 2019 May 9;9(5):e024932. doi: 10.1136/bmjopen-2018-024932. PMID 31076468
- [Derived] Zeng L, Guo J, Wang J, Zhang Q, Li H, Lin R. Clinical re-evaluation of removing blood stasis therapy in treating acute intracerebral hemorrhage safety and efficacy: a protocol for a randomized, controlled, multicenter study (CRRICH Trial). Springerplus. 2016 Sep 1;5(1):1466. doi: 10.1186/s40064-016-3136-y. eCollection 2016. PMID 27652041